CLINICAL TRIAL: NCT02869282
Title: Study Of The Expression Of Circulating And Intra-Tumoral Chemokines In Patients With Prostate Cancer
Brief Title: Circulating And Intra-Tumoral Chemokines In Patients With Prostate Cancer
Acronym: CHEMOPROST
Status: Withdrawn | Type: Observational
Why Stopped: Principal investigator left the study center and nobody took over the study.
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB2011-CHEMOPROST
Record Dates: First submitted 2016-06-28; First posted 2016-08-16 (Estimated); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Additional blood and urine samples (8 ml blood and 20 ml urine tubes)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective cohort: Levels of CXCL1, CCL5, CXCL8 and CXCL12 chemokines and of IL-6 cytokine by ELISA or Luminex technology.
  Interventions: Other: Blood samples; Other: Urine samples

INTERVENTIONS:
Other: Blood samples — Additional blood samples at baseline, 6, 12, 18 and 24 months.
Other: Urine samples — Additional urine samples at baseline, 6, 12, 18 and 24 months.

SUMMARY:
Multicentric, observational, prospective, non-interventional study with occasional biological sample collection (serum bank, urine bank and tumor bank)

DETAILED DESCRIPTION:
This project is an exploratory study, based on the hypothesis of involvement of chemokines in hormonal escape of prostate cancers.

The two main objectives are:

* To describe the variations in expression of chemokines in serum and urine level in patients with prostate cancer
* And to study the disease stage and intra-prostatic concentrations of chemokines based on serum and urine concentrations of chemokines before treatment initiation.

These estimates can be used in future trials set up for the management of prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with a localized or metastatic prostate adenocarcinoma for which a new treatment will be implemented (hormone therapy for single biological relapse or relapses and metastatic hormone-sensitive) or chemotherapy (for biological relapses and / or metastatic hormone-resistant)
* Patients with a detectable PSA (Prostate-Specific Antigen)
* Patients who signed an informed consent
* Patients over 18 years
* Patients belonging to the social security scheme

Exclusion Criteria:

* Active Hepatitis B or C virus
* HIV positive
* Patients who have received prior chemotherapy
* Patients with a second neoplasia treated in the last 5 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a localized or metastatic prostate adenocarcinoma
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Concentration of chemokines initially detectable in the blood or urine and evolution during follow-up: CXCL1, CXCL5, CXCL8, CXCL12, cytokine IL-6. Measurement was made by Luminex or elisa technical | At baseline
Concentration of chemokines initially detectable in the blood or urine and evolution during follow-up: CXCL1, CXCL5, CXCL8, CXCL12, cytokine IL-6. Measurement was made by Luminex or elisa technical | At 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No